CLINICAL TRIAL: NCT04467697
Title: A 6 Month, Open Label, Ambulatory Blood Pressure Monitoring (ABPM) Extension Study
Brief Title: Ambulatory Blood Pressure Monitoring (ABPM) Extension Study of Oral Testosterone Undecanoate in Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marius Pharmaceuticals (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRS-TU-2019EXT
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOV2012-F1-treated (Experimental): Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg in the morning and 400 mg in the evening) or titrated down to a minimum of 100 mg SOV2012-F1 per day (100 mg in the morning) based on plasma T after 14 and 42 days of treatment, intermediate dose levels include total daily doses of 600 mg, 400 mg and 200 mg.
  Interventions: Drug: SOV2012-F1

INTERVENTIONS:
Drug: SOV2012-F1 — Oral preparation of testosterone undecanoate (TU). Strengths of 100 mg TU, 150 mg TU and 200 mg TU

SUMMARY:
The purpose of this six-month treatment study is

* to assess feasibility of a lower starting dose of SOV2012-F1 (daily dose of 400 mg [200 mg with breakfast meal and 200mg with dinner meal]) to titrate individual doses to further enhance efficacy and safety.
* To examine the blood pressure (BP) effects of Marius's oral testosterone undecanoate formulation, SOV2012-F1, using 24-hour ambulatory blood pressure monitoring (ABPM).

DETAILED DESCRIPTION:
This is the six-month treatment extension of Study MRS-TU-2019, which like Study MRS-TU-2019 (NCT03198728), is an open-label study. The MRS-TU-2019 ABPM Extension Study (MRS-TU-2019EXT; NCT04467697), will extend the participation for up to 170 MRS-TU-2019 subjects and to new subjects, for a target of 135 evaluable subjects reaching the 4-month ABPM assessment. All subjects were washed out from previous testosterone therapy if they were not naïve. The study used ABPM monitoring to assess baseline and change from baseline after 120 and 180 days of treatment. The percentage of participants within the normal range for testosterone was assessed after two titration cycles and a total of 90 days of treatment.

ELIGIBILITY:
For all subjects participating in MRS-TU-2019EXT, whether rolling over from MRS-TU-2019 (after washout) or newly enrolling, the following MRS-TU-2019EXT Inclusion/Exclusion Criteria apply:

Inclusion Criteria:

1. Completion of MRS-TU-2019 Day 365/ End of Treatment

Exclusion Criteria:

1. Upper arm circumference > 45 cm.
2. Long distance driving or planned driving trip (> 60 mins duration where the subject is doing the driving) during period of wearing ABPM cuff.
3. Expected / known forthcoming change to antihypertensive medication(s) during the MRS-TU-2019 EXT extension study.
4. Cardiac arrhythmias that, in the opinion of the investigator, interfere with the ability of the ABPM recorder to obtain reliable measurements.
5. Use of T implantable pellets since completion of Day 365/EOT visit in MRS-TU- 2019.

For newly enrolling subjects into MRS-TU-2019EXT (naïve to MRS-TU-2019), the applicable Inclusion/Exclusion criteria from the MRS-TU-2019 study, also must be met :

MRS-TU-2019 Key Inclusion Criteria:

1. Male aged 18 to 65 years, inclusive, at the time of providing informed consent to participate in the study.
2. Hypogonadism defined as having 2 consecutive serum total T levels ≤ 281 ng/dL based on a blood sample, drawn at least 3 days apart, between 7 a.m. and 10 a.m.
3. At least 1 clinical feature consistent with male hypogonadism. If a subject is receiving commercial TRT prior to Screening Visit 1, he must have a history of at least 1 clinical feature consistent with male hypogonadism.
4. Must be naïve to androgen replacement therapy or washed out adequately of prior androgen replacement therapies; willing to cease current T treatment; or currently not taking any T treatment. Subjects must remain off all forms of T, except for dispensed study drug, throughout the entire study.
5. No unstable ongoing concomitant medical conditions. Treated and well-controlled conditions such as type 2 diabetes, hypertension, or dyslipidemia are acceptable with stable medication in place for at least 3 months prior to study entry:

   1. Hemoglobin A1c < 8.0%
   2. BP < 150/90 mm Hg

      * *for MRS-TU-2019EXT ABPM Extension Study, the in-clinic, average BP must be < 140/90 for inclusion into the MRS-TU-2019EXT study.
   3. Low-density lipoprotein cholesterol < 190 mg/dL.
6. Subjects with an endocrine disorder requiring treatment other than hypogonadism must be on a stable dose of replacement medication for at least 3 months prior to study entry.
7. Adequate venous access to allow collection of a number of blood samples via a venous cannula.
8. Written informed consent to participate in the study and ability to comply with all study requirements.

MRS-TU-2019 Key Exclusion Criteria:

1. Serum PSA > 2.5 ng/ml and/or abnormal prostate gland on palpation, e.g., palpable nodes, at Screening Visit 2.
2. Received oral, topical, intranasal, or buccal T therapy within the previous 2 weeks, intramuscular T injection of short-acting duration within the previous 4 weeks, intramuscular T injection of long-acting duration within the previous 20 weeks, or T implantable pellets within the previous 6 months.

   *For ABPM Extension Study Only: Newly Enrolled Subjects to MRS-TU-2019EXT ABPM Extension Study, patients must not have received prior testosterone replacement therapy within 8 weeks of the start of the study, with the exception of T implantable pellets which are excluded for 6 months.
3. Use of any drug that could interfere with measurement or assessment of serum androgen levels, including 5 alpha-reductase inhibitors, anabolic steroids, and drugs with antiandrogenic properties (e.g., spironolactone, cimetidine, flutamide, bicalutamide, and ketoconazole). These drugs must be stopped for at least 1 month prior to study entry (6 months in the case of dutasteride). Patients taking potent, long- acting opiate therapy on a daily basis are not eligible for the study. Conversely, ad hoc use of potent, short-acting opiates for a period of less than 7 days may be permitted after discussion with the Marius Pharmaceuticals medical monitor.
4. Use of over-the-counter products, including natural health products (e.g., food supplements and herbal supplements such as saw palmetto or phytoestrogens) that may affect total T levels, within 7 days prior to study entry.
5. History of drug or alcohol abuse within the past 2 years that in the opinion of the investigator could interfere with study participation and/or influence study efficacy and safety endpoints assessments.
6. Unstable or chronic disease that could interfere with participation in the study or patient safety, including psychiatric disorders.
7. Myocardial infarction, coronary artery surgery, heart failure, stroke, unstable angina, or other unstable cardiovascular disease within the past 6 months.
8. Abnormal ECG considered clinically significant by investigator at Screening.
9. Diagnosis of any cancer within the previous 5 years other than basal or squamous cell skin cancer with clear margins.
10. Any surgical or medical condition that might alter administration of the study drug or comparator, including history of gastric surgery, cholecystectomy, vagotomy, small bowel resection, or any surgical procedure or medications (e.g., GLP-1 agonists and motility agents such as domperidone, metoclopramide, etc.) that might interfere with gastrointestinal motility, pH, or absorption of TU.
11. Duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to screening.
12. Chronic skin conditions on the chest or upper arms that would prevent administration of AndroGel in a manner designed to ensure reliable and consistent absorption thereof
13. Human immunodeficiency virus (HIV) infection.
14. Chronic hepatitis B virus and/or hepatitis C virus (HCV) infection (as determined by positive testing for hepatitis B virus surface antigen or HCV antibody with confirmatory testing, i.e., detectable serum HCV ribonucleic acid [RNA])
15. Clinically significant abnormal laboratory values at screening including but not limited to:

    1. Elevated liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT] > 2X upper limit of normal)
    2. Estimated glomerular filtration rate < 60 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease formula
    3. Hemoglobin < 11.0 g/dL or > 16.0 g/dL. For a subject previously on testosterone replacement therapy with less than 30 days washout prior to screening Visit 2, hemoglobin < 11.0 g/dL or > 17.0 g/dL.
16. Severe or untreated obstructive sleep apnea syndrome.
17. Severe lower urinary tract symptoms (American Urological Association/ IPSS ≥ 19).
18. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study entry.
19. Past, current, or suspected prostate or breast cancer.
20. History of long QT syndrome or unexplained sudden death in a first-degree relative (parent, sibling, or child).
21. Concurrent treatment with medications that may impact the absorption, distribution, metabolism, or excretion of TU or place the subject at risk for treatment with T.
22. Subject has a partner who is currently pregnant or planning pregnancy during the course of the study.
23. Treatment with any other investigational drug within 30 days of study entry or > 5 half- lives (whichever is longer) and at any time during the study.
24. History of noncompliance to medical regimens or potential unreliability in the opinion of the investigator.
25. Unwilling or unable to comply to the dietary requirements for this study.
26. History of polycythemia, either idiopathic or associated with TRT.
27. Donated blood (≥ 500 mL) within the 12-week period prior to study entry.
28. History of an abnormal bleeding tendency or thrombophlebitis within the previous 2 years that is not linked to venipuncture or intravenous cannulation.
29. Onset of gynecomastia within the previous 6 months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 155 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Smith, MB, ChB, Study Director — Syneos Health; Om Dhingra, PhD, Study Chair — Marius Pharmaceuticals
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Coastal Clinic Research Inc, Mobile, Alabama
  - South Florida Medical Research, Aventura, Florida
  - PAB Clinical Research, Brandon, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - My Community Research Center, Miami, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Meridien Research, St. Petersburg, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, PLLC, New York, New York
  - Rapha Institute for Clinical Research, Fayetteville, North Carolina
  - Urologic Consultant of SE Pennyslvania, Bala-Cynwyd, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - University Diabetes Endocrine Consultants, Chattanooga, Tennessee
  - Centex Studies, Inc., Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernstein JS, Dhingra OP. A phase III, single-arm, 6-month trial of a wide-dose range oral testosterone undecanoate product. Ther Adv Urol. 2024 Apr 10;16:17562872241241864. doi: 10.1177/17562872241241864. eCollection 2024 Jan-Dec. PMID 38606384
- See also: MRS-TU-2019 protocol, ClinicalTrials.gov ID: NCT03198728 — https://clinicaltrials.gov/ct2/show/NCT03198728

RESULTS

PARTICIPANT FLOW:
Groups:
- SOV2012-F1-treated: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg in the morning with morning meal and 400 mg in the evening with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 mg twice daily) or 800 mg (400 mg twice daily). All doses taken with meals. Doses were up-titrated at Days 28 and 56 if the measured T-concentration in a NaF/EDTA plasma sample was below 400 ng/dL; down-titrated if the T-concentration was above 900 ng/dL, and no change if between those thresholds.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
Period: Overall Study
Arm/Group | SOV2012-F1-treated
Started | 155
Completed | 135
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 119
  More than one race | 0
  Unknown or Not Reported | 2
Weight at Baseline [Count of Participants; unit: Participants]
  <= 93 kg | 59
  > 93 kg | 96
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.95 (7.343)
Assigned breakfast diet [Count of Participants; unit: Participants]
  Low-fat breakfast | 13
  Normal-fat breakfast | 53
  High-fat breakfast | 80
  Missing | 9
Diabetic Status [Count of Participants; unit: Participants]
  With Diabetes Mellitus | 34
  Without Diabetes Mellitus | 121
Hypertensive Status [Count of Participants; unit: Participants]
  Hypertensive | 96
  Not hypertensive | 56
  Missing | 3
Hypertensive Treatment Status [Count of Participants; unit: Participants]
  With Antihypertensive Therapy at Visit 7E (Day 1 E) | 56
  Without Antihypertensive Therapy at Visit 7E (Day 1 E) | 99
Hypogonadal Status [Count of Participants; unit: Participants]
  Primary | 8
  Secondary | 147

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Average Ambulatory Systolic Blood Pressure After 120 Days Treatment
Description: Change from baseline in 24-hour Ambulatory Systolic Blood Pressure (sBP) after approximately 120 days treatment (Mixed Model Repeated Measures analysis).
Time Frame: 120 days
Population: Extension Treated Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- SOV2012-F1-treated: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg in the morning with morning meal and 400 mg in the evening with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 mg twice daily) or 800 mg (400 mg twice daily). All doses taken with meals.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 139
mmHg
  Baseline | 128.9 [126.8 to 131.0]
  Observed Visit 14E - Day 120E | 130.6 [128.5 to 132.7]
  Change from baseline (Visit 14E - Day 120E) | 1.7 [0.3 to 3.1]

2. Primary Outcome: Plasma and Serum Testosterone Efficacy of Oral SOV2012-F1 With up and Down Titration
Description: Percentage of SOV2012-F1-treated subjects with a plasma NaF/EDTA plasma testosterone (T) Cavg within the normal range after 90 days of treatment using up- and down-titration as appropriate. Measured by Plasma T concentration using a starting daily dose of 400 mg SOV2012-F1.
Time Frame: 90 days
Population: Modified Extension Treated Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- NaF/EDTA PLASMA: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg with morning meal and 400 mg with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 me twice daily) or 800 mg (400 mg twice daily). All doses taken with meals.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
  Patients (n=16) from a single clinical site were excluded from PK-based outcomes due to sample handling errors.
- SERUM: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg with morning meal and 400 mg with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 me twice daily) or 800 mg (400 mg twice daily). All doses taken with meals.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
  Patients (n=16) from a single clinical site were excluded from PK-based outcomes due to sample handling errors.
  Patients were enrolled in the serum sub study.
Arm/Group | NaF/EDTA PLASMA | SERUM
Number analyzed (Participants) | 139 | 89
percentage of participants
  Worst case scenario | 87.8 [82.3 to 93.2] | 86.5 [79.4 to 93.6]
  Day 90 completers: number analyzed (Participants) | 127 | 88
  Day 90 completers | 96.1 [92.7 to 99.4] | 87.5 [80.6 to 94.4]

3. Secondary Outcome: Change From Baseline in 24-hour Average Ambulatory Systolic Blood Pressure After 180 Days Treatment.
Description: Ambulatory Blood Pressure Monitoring (ABPM) of the change from baseline in 24-hour average systolic blood pressure (sBP) after 120 and 180 (+/-) 3 days of treatment (Mixed Model Repeated Measures analysis).
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 139
mmHg
  Baseline | 128.9 [126.8 to 131.0]
  Observed Visit 14E (Day 120E) | 130.6 [128.5 to 132.7]
  Change from baseline (Day 120E - Day 1E) | 1.7 [0.3 to 3.1]
  Observed Visit 16E (Day 180E) | 130.7 [128.6 to 132.8]
  Change from baseline (Day 180E - Day 1E) | 1.8 [0.3 to 3.2]

4. Secondary Outcome: Change From Baseline in 24-hour Average Ambulatory Diastolic Blood Pressure (dBP) After 120 Days and 180 Days of SOV2012-F1 Treatment.
Description: Ambulatory Blood Pressure Monitoring (ABPM) of the change from baseline in 24-hour average diastolic blood pressure (dBP) after 120 Days (+/-) and 180 (+/-) 3 days of treatment (Mixed Model Repeated Measures analysis).
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 139
mmHg
  Baseline | 76.2 [74.6 to 77.9]
  Observed Visit 14E (Day 120E) | 76.9 [75.3 to 78.5]
  Change from Baseline to Visit 14E (Day 120E) | 0.6 [-0.3 to 1.6]
  Observed Visit 16E (Day 180E) | 76.9 [75.2 to 78.5]
  Change from Baseline to Visit 16E (Day 180E) | 0.6 [-0.4 to 1.6]

5. Secondary Outcome: Change From Baseline in 24-hour Average Ambulatory Heart Rate After 120 Days and 180 Days of Treatment.
Description: Ambulatory Blood Pressure Monitoring (ABPM) at 120 Days (+/-3) and after 180 Days (+/- 3) of SOV2012-F1 Treatment (Mixed Model Repeated Measures analysis.
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 139
bpm
  Baseline | 76.3 [74.4 to 78.3]
  Observed Visit 14E (Day 120E) | 77.0 [75.1 to 79.0]
  Change from baseline to Visit 14E (Day 120E) | 0.7 [-0.5 to 1.9]
  Observed Visit 16E (Day 180E) | 78.2 [76.2 to 80.2]
  Change from baseline to Visit 16E (Day 180E) | 1.9 [0.6 to 3.1]

6. Secondary Outcome: Observed and Change From Baseline in Ambulatory Half Hourly Systolic Blood Pressure, After 120 Days and After 180 Days of SOV2012-F1 Treatment.
Description: Observed and change from baseline in Ambulatory half hourly systolic blood pressure as measured by ABPM after 120 Days (+/-3) and after 180 Days (+/-3) of SOV2012-F1 treatment.
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SOV2012-F1-treated - Systolic Blood Pressure (sBP), Baseline: Baseline Ambulatory Blood Pressure Monitoring, sBP.
- SOV2012-F1-treated - Systolic Blood Pressure (sBP), Visit 14E - Day 120E: Observed Ambulatory Blood Pressure Monitoring sBP after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Systolic Blood Pressure (sBP), Change From Baseline, Visit 14E - Day 120E: Change from baseline for Ambulatory Blood Pressure Monitoring sBP after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Systolic Blood Pressure (sBP), Visit 16E - Day 180E: Observed Ambulatory Blood Pressure Monitoring sBP after 180 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Systolic Blood Pressure (sBP), Change From Baseline, Visit 16E - Day 180E: Change from baseline for Ambulatory Blood Pressure Monitoring sBP after 180 days of treatment with SOV2012-F1.
Arm/Group | SOV2012-F1-treated - Systolic Blood Pressure (sBP), Baseline | SOV2012-F1-treated - Systolic Blood Pressure (sBP), Visit 14E - Day 120E | SOV2012-F1-treated - Systolic Blood Pressure (sBP), Change From Baseline, Visit 14E - Day 120E | SOV2012-F1-treated - Systolic Blood Pressure (sBP), Visit 16E - Day 180E | SOV2012-F1-treated - Systolic Blood Pressure (sBP), Change From Baseline, Visit 16E - Day 180E
Number analyzed (Participants) | 155 | 155 | 155 | 155 | 155
mmHg
  0 hours: number analyzed (Participants) | 153 | 136 | 136 | 125 | 125
  0 hours | 133.3 (12.02) | 133.7 (12.90) | 0.7 (13.90) | 133.1 (11.95) | -0.0 (13.17)
  0.5 hours: number analyzed (Participants) | 142 | 120 | 111 | 115 | 109
  0.5 hours | 135.6 (15.23) | 134.2 (13.87) | -0.6 (13.70) | 133.1 (12.22) | -2.2 (15.53)
  1 hour: number analyzed (Participants) | 144 | 125 | 118 | 112 | 106
  1 hour | 133.9 (15.28) | 133.9 (13.53) | 0.4 (15.54) | 135.5 (13.07) | 1.7 (16.52)
  1.5 hours: number analyzed (Participants) | 143 | 128 | 120 | 116 | 109
  1.5 hours | 132.3 (15.32) | 132.8 (13.76) | 0.9 (14.80) | 133.5 (13.75) | 1.6 (16.49)
  2 hours: number analyzed (Participants) | 148 | 131 | 126 | 119 | 117
  2 hours | 131.9 (15.60) | 132.7 (14.17) | 1.9 (16.23) | 132.6 (15.87) | 1.7 (18.07)
  2.5 hours: number analyzed (Participants) | 144 | 127 | 121 | 123 | 118
  2.5 hours | 130.9 (15.29) | 132.6 (15.86) | 1.8 (16.23) | 132.5 (14.08) | 2.4 (16.15)
  3 hours: number analyzed (Participants) | 152 | 127 | 126 | 121 | 121
  3 hours | 130.9 (15.84) | 131.2 (15.86) | 1.0 (18.59) | 132.2 (14.62) | 1.9 (19.28)
  3.5 hours: number analyzed (Participants) | 147 | 129 | 125 | 124 | 119
  3.5 hours | 130.6 (15.54) | 131.5 (16.28) | 1.0 (18.33) | 131.5 (16.53) | 2.0 (17.44)
  4 hours: number analyzed (Participants) | 144 | 133 | 125 | 116 | 109
  4 hours | 130.7 (14.42) | 133.2 (15.35) | 2.2 (14.82) | 131.9 (15.72) | 2.3 (14.91)
  4.5 hours: number analyzed (Participants) | 145 | 131 | 124 | 121 | 117
  4.5 hours | 130.5 (15.73) | 131.5 (15.78) | 1.0 (15.69) | 132.4 (14.70) | 2.6 (15.20)
  5 hours: number analyzed (Participants) | 149 | 129 | 125 | 119 | 116
  5 hours | 129.3 (15.69) | 133.5 (16.69) | 4.8 (17.57) | 130.8 (15.98) | 2.2 (16.13)
  5.5 hours: number analyzed (Participants) | 150 | 129 | 128 | 123 | 121
  5.5 hours | 130.8 (16.20) | 133.8 (16.34) | 3.4 (18.06) | 132.4 (16.83) | 2.5 (17.31)
  6 hours: number analyzed (Participants) | 149 | 130 | 128 | 123 | 120
  6 hours | 130.9 (16.68) | 133.2 (14.86) | 3.2 (16.16) | 132.2 (16.08) | 2.5 (17.79)
  6.5 hours: number analyzed (Participants) | 146 | 132 | 126 | 118 | 112
  6.5 hours | 131.2 (17.44) | 132.4 (15.72) | 2.1 (19.08) | 131.4 (16.31) | 1.6 (19.24)
  7 hours: number analyzed (Participants) | 149 | 134 | 131 | 122 | 120
  7 hours | 131.8 (16.52) | 133.0 (16.16) | 1.3 (17.51) | 129.7 (15.41) | -0.9 (16.11)
  7.5 hours: number analyzed (Participants) | 148 | 130 | 127 | 122 | 119
  7.5 hours | 131.5 (17.07) | 133.3 (15.53) | 1.6 (17.44) | 132.2 (13.53) | 1.2 (17.22)
  8 hours: number analyzed (Participants) | 150 | 132 | 131 | 123 | 121
  8 hours | 132.6 (15.63) | 132.3 (13.22) | -0.8 (16.38) | 131.9 (13.98) | -0.2 (15.65)
  8.5 hours: number analyzed (Participants) | 147 | 127 | 123 | 122 | 118
  8.5 hours | 133.6 (15.24) | 133.7 (14.74) | 0.7 (16.51) | 131.2 (13.51) | -1.4 (14.26)
  9 hours: number analyzed (Participants) | 148 | 127 | 123 | 117 | 114
  9 hours | 133.7 (15.37) | 134.0 (15.99) | 0.6 (16.46) | 131.4 (14.44) | -1.4 (16.61)
  9.5 hours: number analyzed (Participants) | 149 | 128 | 126 | 118 | 118
  9.5 hours | 133.0 (16.47) | 134.7 (15.24) | 1.5 (17.82) | 131.8 (15.67) | -0.4 (15.64)
  10 hours: number analyzed (Participants) | 148 | 129 | 126 | 118 | 114
  10 hours | 132.5 (16.52) | 133.6 (15.09) | 1.4 (17.78) | 134.2 (15.35) | 1.6 (18.16)
  10.5 hours: number analyzed (Participants) | 147 | 129 | 124 | 120 | 115
  10.5 hours | 133.3 (16.54) | 134.9 (17.51) | 1.5 (18.15) | 133.0 (13.51) | -0.3 (16.86)
  11 hours: number analyzed (Participants) | 146 | 132 | 127 | 121 | 116
  11 hours | 132.1 (15.55) | 134.9 (15.43) | 2.6 (16.27) | 132.0 (13.45) | 0.7 (16.09)
  11.5 hours: number analyzed (Participants) | 149 | 127 | 124 | 121 | 119
  11.5 hours | 131.4 (15.99) | 133.5 (14.61) | 1.9 (16.23) | 132.7 (14.42) | 1.7 (15.13)
  12 hours: number analyzed (Participants) | 152 | 133 | 132 | 122 | 122
  12 hours | 129.8 (15.25) | 132.6 (15.45) | 2.7 (16.85) | 131.7 (14.92) | 2.7 (18.01)
  12.5 hours: number analyzed (Participants) | 152 | 132 | 131 | 121 | 120
  12.5 hours | 129.5 (15.29) | 131.4 (15.81) | 2.4 (18.09) | 131.7 (14.19) | 3.4 (16.25)
  13 hours: number analyzed (Participants) | 151 | 132 | 130 | 120 | 119
  13 hours | 126.9 (16.11) | 131.4 (16.17) | 5.3 (17.42) | 130.9 (16.12) | 5.3 (18.77)
  13.5 hours: number analyzed (Participants) | 147 | 133 | 127 | 124 | 120
  13.5 hours | 126.7 (15.55) | 130.1 (17.21) | 3.3 (18.80) | 131.0 (16.29) | 4.6 (18.61)
  14 hours: number analyzed (Participants) | 152 | 134 | 134 | 122 | 122
  14 hours | 125.1 (16.69) | 127.8 (15.68) | 2.9 (18.06) | 128.0 (16.68) | 2.8 (20.12)
  14.5 hours: number analyzed (Participants) | 152 | 134 | 133 | 121 | 120
  14.5 hours | 123.7 (16.27) | 127.2 (16.38) | 3.2 (17.49) | 126.7 (16.22) | 3.4 (19.46)
  15 hours: number analyzed (Participants) | 146 | 133 | 126 | 122 | 116
  15 hours | 122.4 (15.78) | 125.7 (16.48) | 3.5 (18.12) | 127.1 (17.74) | 4.3 (16.45)
  15.5 hours: number analyzed (Participants) | 151 | 133 | 131 | 122 | 120
  15.5 hours | 121.1 (16.98) | 124.2 (16.92) | 3.1 (18.83) | 125.4 (18.38) | 3.6 (20.19)
  16 hours: number analyzed (Participants) | 151 | 135 | 133 | 120 | 118
  16 hours | 119.2 (16.09) | 122.0 (15.24) | 2.3 (17.88) | 123.4 (14.40) | 3.8 (15.77)
  16.5 hours: number analyzed (Participants) | 151 | 134 | 132 | 123 | 121
  16.5 hours | 116.8 (16.02) | 120.5 (16.58) | 3.9 (16.94) | 121.4 (14.99) | 4.5 (17.09)
  17 hours: number analyzed (Participants) | 152 | 134 | 133 | 119 | 118
  17 hours | 116.9 (15.07) | 118.4 (16.39) | 1.0 (17.28) | 120.7 (16.51) | 3.3 (17.81)
  17.5 hours: number analyzed (Participants) | 153 | 133 | 133 | 121 | 121
  17.5 hours | 117.4 (15.03) | 118.4 (16.00) | 0.5 (16.84) | 119.8 (16.35) | 2.1 (15.50)
  18 hours: number analyzed (Participants) | 153 | 133 | 133 | 123 | 123
  18 hours | 116.4 (15.44) | 118.0 (16.12) | 1.3 (17.87) | 118.6 (15.26) | 2.6 (17.10)
  18.5 hours: number analyzed (Participants) | 149 | 131 | 127 | 123 | 119
  18.5 hours | 117.7 (15.18) | 117.4 (16.31) | 0.1 (16.51) | 118.5 (15.02) | 2.3 (15.92)
  19 hours: number analyzed (Participants) | 151 | 135 | 133 | 122 | 120
  19 hours | 116.1 (14.22) | 117.2 (15.37) | 1.1 (16.02) | 118.1 (16.61) | 1.9 (16.23)
  19.5 hours: number analyzed (Participants) | 149 | 133 | 129 | 123 | 120
  19.5 hours | 116.5 (15.54) | 118.5 (15.24) | 2.4 (16.40) | 117.9 (16.19) | 2.0 (16.59)
  20 hours: number analyzed (Participants) | 149 | 135 | 134 | 121 | 120
  20 hours | 117.4 (16.25) | 117.7 (16.48) | 0.6 (16.77) | 119.0 (15.33) | 1.1 (14.78)
  20.5 hours: number analyzed (Participants) | 148 | 134 | 130 | 120 | 117
  20.5 hours | 118.2 (16.81) | 117.9 (16.29) | 0.4 (18.78) | 120.2 (17.50) | 1.9 (16.49)
  21 hours: number analyzed (Participants) | 150 | 128 | 126 | 122 | 120
  21 hours | 118.4 (15.85) | 120.7 (16.36) | 1.7 (19.28) | 121.2 (16.42) | 2.0 (17.72)
  21.5 hours: number analyzed (Participants) | 150 | 131 | 129 | 155 | 122
  21.5 hours | 123.0 (15.13) | 121.8 (16.57) | -1.1 (17.92) | 124.7 (16.86) | 1.9 (17.95)
  22 hours: number analyzed (Participants) | 143 | 124 | 118 | 117 | 110
  22 hours | 123.8 (16.88) | 124.1 (15.37) | 0.9 (18.73) | 126.0 (15.12) | 3.2 (17.04)
  22.5 hours: number analyzed (Participants) | 139 | 120 | 109 | 109 | 100
  22.5 hours | 127.1 (17.61) | 129.5 (15.39) | 3.3 (17.35) | 128.3 (16.56) | 4.6 (16.98)
  23 hours: number analyzed (Participants) | 133 | 116 | 99 | 110 | 96
  23 hours | 129.1 (16.44) | 129.4 (15.25) | 0.4 (17.41) | 132.6 (15.73) | 4.8 (16.49)
  23.5 hours: number analyzed (Participants) | 130 | 122 | 103 | 111 | 97
  23.5 hours | 131.0 (13.83) | 130.4 (13.41) | -0.9 (13.66) | 131.6 (14.62) | 0.9 (15.08)

7. Secondary Outcome: Observed and Change From Baseline in Ambulatory Half Hourly Diastolic Blood Pressure, After 120 Days and After 180 Days of SOV2012-F1 Treatment.
Description: Observed and change from baseline in Ambulatory half hourly diastolic blood pressure as measured by ABPM after 120 Days (+/-3) and after 180 Days (+/-3) of SOV2012-F1 treatment.
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Baseline: Baseline Ambulatory Blood Pressure Monitoring, dBP.
- SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Visit 14E - Day 120E: Observed Ambulatory Blood Pressure Monitoring dBP after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Change From Baseline, Visit 14E - Day 120E: Change from baseline for Ambulatory Blood Pressure Monitoring dBP after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Visit 16E - Day 180E: Observed Ambulatory Blood Pressure Monitoring dBP after 180 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Change From Baseline, Visit 16E - Day 180E: Change from baseline for Ambulatory Bood Pressure Monitoring dBP after 180 days of treatment with SOV2012-F1.
Arm/Group | SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Baseline | SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Visit 14E - Day 120E | SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Change From Baseline, Visit 14E - Day 120E | SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Visit 16E - Day 180E | SOV2012-F1-treated - Diastolic Blood Pressure (dBP), Change From Baseline, Visit 16E - Day 180E
Number analyzed (Participants) | 155 | 155 | 155 | 155 | 155
mmHg
  0 hours: number analyzed (Participants) | 153 | 136 | 136 | 125 | 125
  0 hours | 83.7 (9.78) | 83.9 (10.09) | 0.6 (9.90) | 83.3 (9.16) | 0.1 (9.51)
  0.5 hours: number analyzed (Participants) | 142 | 120 | 111 | 115 | 109
  0.5 hours | 83.5 (11.71) | 82.2 (10.36) | -1.0 (11.35) | 82.9 (10.30) | -0.2 (11.42)
  1 hour: number analyzed (Participants) | 144 | 125 | 118 | 112 | 106
  1 hour | 81.7 (11.42) | 82.0 (11.10) | 0.3 (12.69) | 82.9 (11.19) | 1.4 (12.38)
  1.5 hours: number analyzed (Participants) | 143 | 128 | 120 | 116 | 109
  1.5 hours | 80.9 (12.37) | 80.8 (10.80) | 0.6 (10.81) | 81.1 (10.97) | 1.2 (12.32)
  2 hours: number analyzed (Participants) | 148 | 131 | 126 | 119 | 117
  2 hours | 81.2 (11.66) | 80.4 (12.83) | 0.4 (12.91) | 79.8 (10.62) | -0.0 (12.29)
  2.5 hours: number analyzed (Participants) | 144 | 127 | 121 | 123 | 118
  2.5 hours | 79.0 (11.54) | 79.4 (12.28) | 0.7 (15.36) | 80.2 (11.05) | 1.6 (13.62)
  3 hours: number analyzed (Participants) | 152 | 127 | 126 | 121 | 121
  3 hours | 78.9 (12.13) | 79.0 (12.82) | -0.1 (14.34) | 79.5 (11.60) | 0.5 (14.85)
  3.5 hours: number analyzed (Participants) | 147 | 129 | 125 | 124 | 119
  3.5 hours | 79.8 (12.56) | 79.9 (12.25) | -0.2 (14.17) | 79.1 (11.75) | -0.2 (12.58)
  4 hours: number analyzed (Participants) | 144 | 133 | 125 | 116 | 109
  4 hours | 79.1 (11.36) | 80.7 (11.87) | 1.2 (12.19) | 79.2 (11.17) | 0.5 (10.83)
  4.5 hours: number analyzed (Participants) | 145 | 131 | 124 | 121 | 117
  4.5 hours | 79.6 (12.55) | 79.3 (12.48) | -0.5 (12.84) | 79.3 (10.53) | 0.2 (12.21)
  5 hours: number analyzed (Participants) | 149 | 129 | 125 | 119 | 116
  5 hours | 78.1 (13.51) | 79.9 (12.15) | 2.2 (13.74) | 78.3 (12.22) | 0.9 (12.21)
  5.5 hours: number analyzed (Participants) | 150 | 129 | 128 | 123 | 121
  5.5 hours | 77.8 (12.39) | 80.9 (14.40) | 3.3 (14.05) | 78.9 (12.41) | 1.5 (13.31)
  6 hours: number analyzed (Participants) | 149 | 130 | 128 | 123 | 120
  6 hours | 79.5 (12.94) | 79.5 (12.27) | 0.1 (12.22) | 78.3 (11.47) | -0.5 (13.33)
  6.5 hours: number analyzed (Participants) | 146 | 132 | 126 | 118 | 112
  6.5 hours | 78.5 (12.89) | 78.8 (11.51) | 0.3 (13.18) | 79.1 (12.72) | 1.3 (14.39)
  7 hours: number analyzed (Participants) | 149 | 134 | 131 | 122 | 120
  7 hours | 78.5 (12.96) | 78.9 (11.75) | -0.0 (11.94) | 77.9 (11.92) | 0.3 (12.75)
  7.5 hours: number analyzed (Participants) | 148 | 130 | 127 | 122 | 119
  7.5 hours | 79.5 (13.48) | 79.5 (12.69) | 0.4 (14.08) | 79.2 (11.82) | -0.0 (12.66)
  8 hours: number analyzed (Participants) | 150 | 132 | 131 | 123 | 121
  8 hours | 80.3 (12.73) | 79.2 (11.24) | -1.5 (13.63) | 78.9 (11.10) | -0.7 (12.71)
  8.5 hours: number analyzed (Participants) | 147 | 127 | 123 | 122 | 118
  8.5 hours | 80.1 (12.22) | 80.3 (11.82) | 0.8 (12.80) | 78.9 (10.52) | -0.6 (12.20)
  9 hours: number analyzed (Participants) | 148 | 127 | 123 | 117 | 114
  9 hours | 81.0 (12.64) | 80.6 (12.26) | 0.2 (12.77) | 79.1 (11.75) | -1.6 (13.58)
  9.5 hours: number analyzed (Participants) | 149 | 128 | 126 | 118 | 118
  9.5 hours | 80.3 (13.11) | 80.4 (12.24) | 0.1 (13.46) | 79.8 (11.99) | 0.4 (14.33)
  10 hours: number analyzed (Participants) | 148 | 129 | 126 | 118 | 114
  10 hours | 81.1 (12.61) | 80.5 (11.79) | -0.6 (12.75) | 80.4 (12.45) | -0.5 (13.58)
  10.5 hours: number analyzed (Participants) | 147 | 129 | 124 | 120 | 115
  10.5 hours | 80.4 (12.48) | 79.9 (12.02) | -0.3 (13.59) | 79.8 (11.75) | -0.5 (12.65)
  11 hours: number analyzed (Participants) | 146 | 132 | 127 | 121 | 116
  11 hours | 79.2 (11.71) | 80.0 (12.01) | 0.6 (12.60) | 79.1 (12.60) | 0.2 (13.38)
  11.5 hours: number analyzed (Participants) | 149 | 127 | 124 | 121 | 119
  11.5 hours | 79.1 (12.48) | 79.3 (11.81) | -0.4 (12.44) | 77.7 (12.77) | -0.8 (12.62)
  12 hours: number analyzed (Participants) | 152 | 133 | 132 | 122 | 122
  12 hours | 77.6 (12.75) | 79.8 (11.25) | 1.9 (12.60) | 77.7 (12.12) | 0.1 (14.20)
  12.5 hours: number analyzed (Participants) | 152 | 132 | 131 | 121 | 120
  12.5 hours | 78.3 (13.37) | 78.4 (11.90) | 0.2 (13.96) | 77.5 (11.80) | -0.3 (13.59)
  13 hours: number analyzed (Participants) | 151 | 132 | 130 | 120 | 119
  13 hours | 75.1 (12.71) | 76.9 (12.52) | 2.4 (12.37) | 76.3 (12.20) | 2.3 (13.55)
  13.5 hours: number analyzed (Participants) | 147 | 133 | 127 | 124 | 120
  13.5 hours | 75.0 (12.23) | 76.7 (13.26) | 1.9 (14.89) | 76.2 (11.72) | 1.5 (14.28)
  14 hours: number analyzed (Participants) | 152 | 134 | 134 | 122 | 122
  14 hours | 73.1 (12.93) | 74.4 (11.73) | 1.4 (14.13) | 74.0 (12.41) | 0.6 (15.89)
  14.5 hours: number analyzed (Participants) | 152 | 134 | 133 | 121 | 120
  14.5 hours | 72.3 (12.97) | 74.2 (12.82) | 1.6 (14.56) | 73.0 (11.84) | 1.1 (14.22)
  15 hours: number analyzed (Participants) | 146 | 133 | 126 | 122 | 116
  15 hours | 70.7 (12.39) | 72.5 (12.36) | 2.1 (14.20) | 74.3 (12.43) | 3.8 (13.00)
  15.5 hours: number analyzed (Participants) | 151 | 133 | 131 | 122 | 120
  15.5 hours | 69.8 (13.53) | 71.8 (12.22) | 1.6 (16.12) | 72.5 (13.17) | 2.3 (15.89)
  16 hours: number analyzed (Participants) | 151 | 135 | 133 | 120 | 118
  16 hours | 68.3 (13.06) | 70.5 (12.46) | 1.5 (15.77) | 71.0 (11.59) | 1.9 (13.87)
  16.5 hours: number analyzed (Participants) | 151 | 134 | 132 | 123 | 121
  16.5 hours | 67.7 (12.71) | 69.8 (11.20) | 2.1 (13.03) | 69.9 (12.66) | 2.4 (15.69)
  17 hours: number analyzed (Participants) | 152 | 134 | 133 | 119 | 118
  17 hours | 67.2 (11.77) | 69.1 (12.04) | 1.8 (13.27) | 69.6 (12.38) | 2.6 (14.27)
  17.5 hours: number analyzed (Participants) | 155 | 133 | 133 | 121 | 121
  17.5 hours | 67.6 (11.91) | 69.3 (12.42) | 1.2 (14.70) | 69.0 (12.62) | 0.8 (13.16)
  18 hours: number analyzed (Participants) | 155 | 133 | 133 | 123 | 123
  18 hours | 67.7 (12.63) | 68.9 (11.62) | 0.9 (13.79) | 68.0 (12.20) | 0.5 (14.84)
  18.5 hours: number analyzed (Participants) | 149 | 131 | 127 | 123 | 119
  18.5 hours | 68.3 (11.82) | 68.6 (11.46) | 0.2 (13.77) | 68.4 (12.08) | 0.7 (12.81)
  19 hours: number analyzed (Participants) | 151 | 135 | 133 | 122 | 120
  19 hours | 67.6 (11.78) | 68.3 (11.14) | 0.7 (12.97) | 69.2 (12.48) | 1.2 (12.54)
  19.5 hours: number analyzed (Participants) | 149 | 133 | 129 | 123 | 120
  19.5 hours | 67.9 (11.62) | 69.4 (12.85) | 1.5 (13.41) | 68.9 (13.12) | 1.2 (12.89)
  20 hours: number analyzed (Participants) | 149 | 135 | 134 | 121 | 120
  20 hours | 69.6 (12.43) | 68.5 (12.95) | -1.3 (13.93) | 69.8 (12.88) | -0.4 (13.50)
  20.5 hours: number analyzed (Participants) | 148 | 134 | 130 | 120 | 117
  20.5 hours | 69.8 (13.04) | 68.9 (12.56) | -0.8 (14.42) | 69.9 (13.25) | -0.2 (13.22)
  21 hours: number analyzed (Participants) | 150 | 128 | 126 | 122 | 120
  21 hours | 70.3 (13.04) | 70.8 (13.56) | 0.1 (15.23) | 72.8 (13.05) | 1.9 (14.26)
  21.5 hours: number analyzed (Participants) | 150 | 131 | 129 | 155 | 122
  21.5 hours | 73.8 (13.00) | 72.6 (14.23) | -1.4 (15.16) | 74.8 (13.79) | 1.0 (15.12)
  22 hours: number analyzed (Participants) | 143 | 124 | 118 | 117 | 110
  22 hours | 74.9 (13.38) | 74.3 (13.15) | -0.0 (15.63) | 76.2 (12.44) | 2.4 (13.20)
  22.5 hours: number analyzed (Participants) | 139 | 120 | 109 | 109 | 100
  22.5 hours | 77.8 (13.39) | 80.4 (13.33) | 3.6 (14.74) | 77.5 (12.74) | 2.3 (11.92)
  23 hours: number analyzed (Participants) | 133 | 116 | 99 | 110 | 96
  23 hours | 80.6 (12.53) | 79.3 (13.72) | -0.8 (13.52) | 81.6 (12.13) | 1.7 (12.87)
  23.5 hours: number analyzed (Participants) | 130 | 122 | 103 | 111 | 97
  23.5 hours | 81.8 (11.05) | 82.1 (12.17) | 0.3 (12.82) | 80.6 (10.98) | -0.3 (11.30)

8. Secondary Outcome: Observed and Change From Baseline in Ambulatory Half Hourly Heart Rate Measurement, After 120 Days and After 180 Days (±3) of SOV2012-F1 Treatment.
Description: Observed and change from baseline in Ambulatory half hourly heart rate as measured by ABPM after 120 Days (+/-3) and after 180 Days (+/-3) of SOV2012-F1 treatment.
Time Frame: 120 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- SOV2012-F1-treated - Heart Rate (Bpm), Baseline: Baseline Ambulatory Blood Pressure Monitoring (ABPM) heart rate.
- SOV2012-F1-treated - Heart Rate (Bpm), Visit 14E - Day 120E: Observed Ambulatory Blood Pressure Monitoring heart rate after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Heart Rate (Bpm), Change From Baseline, Visit 14E - Day 120E: Change from Baseline for Ambulatory Blood Pressure Monitoring heart rate after 120 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Heart Rate (Bpm), Visit 16E - Day 180E: Observed Ambulatory Blood Pressure Monitoring heart rate after 180 days of treatment with SOV2012-F1.
- SOV2012-F1-treated - Heart Rate (Bpm), Change From Baseline, Visit 16E - Day 180E: Change from Baseline for Ambulatory Blood Pressure Monitoring heart rate after 180 days of treatment with SOV2012-F1.
Arm/Group | SOV2012-F1-treated - Heart Rate (Bpm), Baseline | SOV2012-F1-treated - Heart Rate (Bpm), Visit 14E - Day 120E | SOV2012-F1-treated - Heart Rate (Bpm), Change From Baseline, Visit 14E - Day 120E | SOV2012-F1-treated - Heart Rate (Bpm), Visit 16E - Day 180E | SOV2012-F1-treated - Heart Rate (Bpm), Change From Baseline, Visit 16E - Day 180E
Number analyzed (Participants) | 155 | 155 | 155 | 155 | 155
bpm
  0 hours: number analyzed (Participants) | 153 | 136 | 136 | 125 | 125
  0 hours | 72.6 (10.22) | 74.5 (10.15) | 2.3 (9.72) | 74.5 (11.63) | 3.0 (10.17)
  0.5 hours: number analyzed (Participants) | 142 | 120 | 111 | 115 | 109
  0.5 hours | 76.0 (12.94) | 77.6 (12.70) | 0.5 (11.06) | 78.1 (14.86) | 3.4 (14.24)
  1 hour: number analyzed (Participants) | 144 | 125 | 118 | 112 | 106
  1 hour | 77.7 (15.77) | 80.4 (13.03) | 2.4 (16.11) | 81.1 (16.17) | 4.5 (18.28)
  1.5 hours: number analyzed (Participants) | 143 | 128 | 120 | 116 | 109
  1.5 hours | 79.9 (12.93) | 80.8 (16.36) | 1.4 (16.77) | 83.1 (14.84) | 3.6 (15.81)
  2 hours: number analyzed (Participants) | 148 | 131 | 126 | 119 | 117
  2 hours | 80.7 (15.79) | 80.8 (13.53) | 0.8 (16.59) | 82.9 (15.78) | 3.6 (16.50)
  2.5 hours: number analyzed (Participants) | 144 | 127 | 121 | 123 | 118
  2.5 hours | 79.4 (14.63) | 80.3 (14.60) | 0.7 (15.94) | 82.8 (15.84) | 4.4 (15.38)
  3 hours: number analyzed (Participants) | 152 | 127 | 126 | 121 | 121
  3 hours | 79.0 (13.08) | 79.5 (13.15) | 0.2 (14.08) | 80.3 (15.85) | 2.7 (14.96)
  3.5 hours: number analyzed (Participants) | 147 | 129 | 125 | 124 | 119
  3.5 hours | 79.3 (15.29) | 80.1 (13.81) | 0.4 (18.50) | 79.9 (16.20) | 2.3 (18.42)
  4 hours: number analyzed (Participants) | 144 | 133 | 125 | 116 | 109
  4 hours | 78.4 (14.73) | 79.7 (14.59) | 1.1 (15.37) | 80.1 (16.23) | 2.8 (18.74)
  4.5 hours: number analyzed (Participants) | 145 | 131 | 124 | 121 | 117
  4.5 hours | 79.1 (15.18) | 79.2 (13.65) | 0.4 (16.29) | 79.9 (15.05) | 3.0 (16.75)
  5 hours: number analyzed (Participants) | 149 | 129 | 125 | 119 | 116
  5 hours | 79.0 (15.42) | 80.5 (14.79) | 1.2 (16.09) | 79.7 (15.39) | 2.9 (14.93)
  5.5 hours: number analyzed (Participants) | 150 | 129 | 128 | 123 | 121
  5.5 hours | 78.5 (14.56) | 80.6 (13.19) | 1.9 (15.36) | 81.0 (16.05) | 4.0 (16.48)
  6 hours: number analyzed (Participants) | 149 | 130 | 128 | 123 | 120
  6 hours | 79.3 (14.41) | 80.5 (13.26) | 1.2 (15.46) | 80.4 (14.02) | 2.9 (15.49)
  6.5 hours: number analyzed (Participants) | 146 | 132 | 126 | 118 | 112
  6.5 hours | 79.2 (15.03) | 80.1 (14.40) | 1.5 (14.90) | 80.4 (13.94) | 3.2 (15.91)
  7 hours: number analyzed (Participants) | 149 | 134 | 131 | 122 | 120
  7 hours | 80.6 (15.04) | 80.9 (13.85) | 0.8 (14.83) | 79.8 (13.27) | 0.6 (15.44)
  7.5 hours: number analyzed (Participants) | 148 | 130 | 127 | 122 | 119
  7.5 hours | 80.0 (14.51) | 79.5 (13.66) | -0.3 (15.20) | 81.1 (14.52) | 2.4 (14.98)
  8 hours: number analyzed (Participants) | 150 | 132 | 131 | 123 | 121
  8 hours | 81.5 (14.63) | 80.8 (14.18) | -0.9 (15.86) | 80.8 (14.34) | 0.5 (15.15)
  8.5 hours: number analyzed (Participants) | 147 | 127 | 123 | 122 | 118
  8.5 hours | 80.0 (14.09) | 79.9 (14.41) | -0.1 (13.89) | 79.9 (13.34) | 0.6 (14.18)
  9 hours: number analyzed (Participants) | 148 | 127 | 123 | 117 | 114
  9 hours | 80.1 (13.86) | 80.9 (14.06) | 0.2 (14.70) | 82.2 (13.93) | 2.5 (15.45)
  9.5 hours: number analyzed (Participants) | 149 | 128 | 126 | 118 | 118
  9.5 hours | 79.9 (14.21) | 80.1 (16.09) | -0.1 (14.18) | 81.8 (13.70) | 2.1 (16.58)
  10 hours: number analyzed (Participants) | 148 | 129 | 126 | 118 | 114
  10 hours | 81.8 (16.28) | 80.6 (15.75) | -1.0 (15.28) | 82.1 (14.95) | 1.1 (16.53)
  10.5 hours: number analyzed (Participants) | 147 | 129 | 124 | 120 | 115
  10.5 hours | 80.4 (14.75) | 78.4 (13.73) | -2.2 (13.59) | 80.7 (13.82) | 1.2 (15.30)
  11 hours: number analyzed (Participants) | 146 | 132 | 127 | 121 | 116
  11 hours | 79.9 (14.07) | 80.5 (15.79) | 0.3 (14.52) | 80.8 (13.14) | 2.0 (13.84)
  11.5 hours: number analyzed (Participants) | 149 | 127 | 124 | 121 | 119
  11.5 hours | 79.8 (14.31) | 79.4 (14.58) | -1.0 (16.26) | 80.2 (15.05) | 0.9 (14.64)
  12 hours: number analyzed (Participants) | 152 | 133 | 132 | 122 | 122
  12 hours | 79.5 (13.80) | 79.3 (15.02) | -0.5 (15.77) | 79.8 (14.57) | 1.2 (13.92)
  12.5 hours: number analyzed (Participants) | 152 | 132 | 131 | 121 | 120
  12.5 hours | 78.8 (13.66) | 79.1 (15.12) | 0.7 (15.81) | 78.9 (14.33) | 0.8 (13.62)
  13 hours: number analyzed (Participants) | 151 | 132 | 130 | 120 | 119
  13 hours | 76.4 (12.04) | 77.6 (13.23) | 1.7 (13.59) | 77.8 (14.49) | 2.3 (14.37)
  13.5 hours: number analyzed (Participants) | 147 | 133 | 127 | 124 | 120
  13.5 hours | 75.8 (12.05) | 77.6 (13.90) | 2.3 (14.01) | 78.1 (15.15) | 3.7 (14.77)
  14 hours: number analyzed (Participants) | 152 | 134 | 134 | 122 | 122
  14 hours | 75.6 (12.47) | 75.5 (13.44) | 0.1 (13.93) | 75.9 (13.63) | 1.0 (13.19)
  14.5 hours: number analyzed (Participants) | 152 | 134 | 133 | 121 | 120
  14.5 hours | 73.3 (12.74) | 75.5 (12.80) | 2.0 (13.70) | 75.1 (13.76) | 2.3 (14.03)
  15 hours: number analyzed (Participants) | 146 | 133 | 126 | 122 | 116
  15 hours | 72.5 (11.47) | 74.5 (12.37) | 2.0 (13.02) | 74.3 (13.49) | 2.3 (11.29)
  15.5 hours: number analyzed (Participants) | 151 | 133 | 131 | 122 | 120
  15.5 hours | 72.0 (12.06) | 73.3 (12.41) | 1.1 (12.61) | 72.9 (12.71) | 1.1 (12.61)
  16 hours: number analyzed (Participants) | 151 | 135 | 133 | 120 | 118
  16 hours | 70.8 (12.21) | 71.9 (12.01) | 1.0 (11.48) | 72.6 (12.32) | 1.7 (12.40)
  16.5 hours: number analyzed (Participants) | 151 | 134 | 132 | 123 | 121
  16.5 hours | 69.5 (10.97) | 71.0 (11.59) | 1.8 (12.13) | 72.0 (13.19) | 2.5 (12.75)
  17 hours: number analyzed (Participants) | 152 | 134 | 133 | 119 | 118
  17 hours | 69.7 (12.03) | 70.5 (11.83) | 0.8 (11.60) | 70.2 (13.07) | 0.8 (12.09)
  17.5 hours: number analyzed (Participants) | 153 | 133 | 133 | 121 | 121
  17.5 hours | 69.5 (10.94) | 69.9 (11.53) | 0.5 (12.57) | 70.3 (13.13) | 0.4 (13.22)
  18 hours: number analyzed (Participants) | 153 | 133 | 133 | 123 | 123
  18 hours | 68.2 (11.40) | 68.7 (10.61) | 0.5 (11.33) | 69.4 (12.94) | 1.4 (12.65)
  18.5 hours: number analyzed (Participants) | 149 | 131 | 127 | 123 | 119
  18.5 hours | 68.4 (11.24) | 68.4 (11.23) | 0.2 (10.66) | 69.5 (13.10) | 1.4 (13.11)
  19 hours: number analyzed (Participants) | 151 | 135 | 133 | 122 | 120
  19 hours | 67.4 (10.88) | 67.6 (10.68) | 0.4 (10.56) | 69.2 (13.04) | 2.1 (11.70)
  19.5 hours: number analyzed (Participants) | 149 | 133 | 129 | 123 | 120
  19.5 hours | 67.1 (11.10) | 67.4 (11.15) | 0.9 (11.08) | 69.8 (12.70) | 2.7 (12.47)
  20 hours: number analyzed (Participants) | 149 | 135 | 134 | 121 | 120
  20 hours | 68.5 (11.67) | 66.8 (10.85) | -1.2 (11.74) | 67.7 (12.50) | -0.4 (13.55)
  20.5 hours: number analyzed (Participants) | 148 | 134 | 130 | 120 | 117
  20.5 hours | 68.5 (12.28) | 67.3 (11.70) | -0.8 (13.57) | 68.4 (12.36) | 0.0 (12.43)
  21 hours: number analyzed (Participants) | 150 | 128 | 126 | 122 | 120
  21 hours | 69.0 (11.22) | 68.1 (12.46) | -0.6 (13.25) | 68.8 (12.70) | -0.2 (12.68)
  21.5 hours: number analyzed (Participants) | 150 | 131 | 129 | 155 | 122
  21.5 hours | 69.9 (13.57) | 68.2 (11.52) | -1.4 (14.26) | 71.6 (13.75) | 1.4 (13.83)
  22 hours: number analyzed (Participants) | 143 | 124 | 118 | 117 | 110
  22 hours | 71.3 (15.14) | 70.4 (13.80) | -0.6 (16.58) | 73.0 (14.46) | 3.1 (14.46)
  22.5 hours: number analyzed (Participants) | 139 | 120 | 109 | 109 | 100
  22.5 hours | 73.6 (12.08) | 75.0 (15.82) | 2.2 (16.44) | 75.3 (16.29) | 3.1 (14.80)
  23 hours: number analyzed (Participants) | 133 | 116 | 99 | 110 | 96
  23 hours | 75.9 (16.45) | 74.5 (13.07) | 1.2 (12.72) | 75.9 (13.58) | 1.8 (12.75)
  23.5 hours: number analyzed (Participants) | 130 | 122 | 103 | 111 | 97
  23.5 hours | 74.2 (11.67) | 77.8 (13.99) | 3.2 (14.69) | 79.6 (17.40) | 3.7 (12.82)

9. Secondary Outcome: Percentage of SOV2012-F1-Treated Subjects With Maximum Plasma Testosterone Concentration After 90 Days of Treatment: < 1.5X Upper Limit of Normal (ULN); 1.8 to ≤ 2.5X ULN; > 2.5X ULN
Description: Percentage of SOV2012-F1 treated subjects with maximum NaF/EDTA plasma T levels falling into three concentration groups after 90 days of treatment with SOV2012-F1.
Time Frame: 90 days
Population: Modified Extension Treatment Set
Measure: Count of Participants; unit: Participants
Arm/Group | NaF/EDTA PLASMA
Number analyzed (Participants) | 139
Participants
  Plasma T Cmax <=1200 ng/dL after 90days: number analyzed (Participants) | 130
  Plasma T Cmax <=1200 ng/dL after 90days | 114
  Plasma T Cmax <=1440 ng/dL to 2000 ng/dL after 90days: number analyzed (Participants) | 130
  Plasma T Cmax <=1440 ng/dL to 2000 ng/dL after 90days | 5
  Plasma T Cmax >2000 ng/dL after 90days: number analyzed (Participants) | 130
  Plasma T Cmax >2000 ng/dL after 90days | 0

10. Secondary Outcome: Percentage of SOV2012-F1-Treated Subjects With Maximum Serum Testosterone Concentration After 90 Days of Treatment: < 1.5X Upper Limit of Normal (ULN); 1.8 to ≤ 2.5X ULN; > 2.5X ULN
Description: Percentage of SOV2012-F1 treated subjects with maximum serum levels falling into three concentration groups after 90 days of treatment with SOV2012-F1.
Time Frame: 90 days
Population: Modified Extension Treatment Set
Measure: Count of Participants; unit: Participants
Groups:
- SERUM: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg with morning meal and 400 mg with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 me twice daily) or 800 mg (400 mg twice daily). All doses taken with meals.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
  Patients (n=16) from a single clinical site were excluded from PK-based outcomes due to sample handling errors.
  Patients were participants in the Serum sub study.
Arm/Group | SERUM
Number analyzed (Participants) | 89
Participants
  T Cmax <=1500 ng/dL After 90 Days | 81
  T Cmax 1800 to 2500 ng/dL After 90 Days | 4
  T Cmax >2500 ng/dL After 90 Days | 0

11. Other Pre Specified Outcome: AEs, SAEs and AEs Leading to MRS-TU-2019EXT Study Withdrawal of SOV2012-F1 Treated Subjects.
Description: Number of subjects of adverse events (AEs), serious adverse events (SAEs), and AEs leading to study withdrawal in SOV2012-F1-treated subjects
Time Frame: 180 days
Population: Extension Treated Set
Measure: Count of Participants; unit: Participants
Arm/Group | SOV2012-F1-treated
Number analyzed (Participants) | 155
Participants
  Any TEAEs | 58
  Any Serious TEAEs | 2
  Any Treatment-related TEAEs | 13
  Any Treatment-related Serious TEAEs | 0
  Any Severe TEAEs | 3
  Any Treatment-related Severe TEAEs | 0
  Any TEAEs leading to Discontinuation from Study Drug | 1
  Any TEAEs leading to Death | 0
  Any MACE | 0
  Any TEAEs of Hypertension or Blood Pressure Increased | 6

12. Other Pre Specified Outcome: Observed and Change From Baseline in Systolic Blood Pressure Using In-clinic Measurement.
Description: Measured by in-clinic BP measurement of sBP, mmHg, observed and change from baseline at baseline, 90, 120 and 180 days after treatment with SOV2012-F1.
Time Frame: Baseline, 90, 119 and 179 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SOV2012-F1-treated, Observed: Observed systolic BP measured in-clinic at baseline, and 90, 120 and 180 days of treatment with SOV2012-F1
- SOV2012-F1-treated, Change From Baseline: Change in baseline for systolic BP measured in-clinic after 90, 120 and 180 days of treatment with SOV2012-F1
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
mmHg
  Baseline EXT: number analyzed (Participants) | 152 | 152
  Baseline EXT | 126.10 (9.800) | 0 (0)
  Visit 12E - Day 90E: number analyzed (Participants) | 146 | 145
  Visit 12E - Day 90E | 127.89 (9.961) | 2.06 (10.303)
  Visit 13E - Day 119E: number analyzed (Participants) | 141 | 140
  Visit 13E - Day 119E | 128.51 (10.912) | 2.70 (10.695)
  Visit 15E - Day 179E: number analyzed (Participants) | 132 | 131
  Visit 15E - Day 179E | 128.09 (10.012) | 2.39 (10.522)

13. Other Pre Specified Outcome: Observed and Change From Baseline in Heartrate (HR) Obtained In-clinic During the Treatment Period.
Description: Measured by in-clinic HR measurement, beats per minute during the treatment period, at baseline, and after 90, 120 and 180 days of treatment with SOV2012-F1.
Time Frame: Baseline, 90, 119 and 179 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: beats/minute
Groups:
- SOV2012-F1-treated, Observed: Observed heartrate (HR) measured in-clinic at baseline, and 90, 120 and 180 days of treatment with SOV2012-F1.
- SOV2012-F1-treated, Change From Baseline: Change from baseline for heartrate (HR) measured in-clinic at 90, 120 and 180 days of treatment with SOV2012-F1.
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
beats/minute
  Baseline EXT | 71.9 (9.48) | 0 (0)
  Visit 12E - Day 90E: number analyzed (Participants) | 146 | 146
  Visit 12E - Day 90E | 73.9 (9.42) | 1.9 (9.09)
  Visit 13E - Day 119E: number analyzed (Participants) | 141 | 141
  Visit 13E - Day 119E | 72.9 (9.40) | 1.1 (9.13)
  Visit 15E - Day 179E: number analyzed (Participants) | 132 | 132
  Visit 15E - Day 179E | 74.3 (10.26) | 2.6 (9.37)

14. Other Pre Specified Outcome: Observed and Change From Baseline in Hematology Parameters in Liver Function Tests of ALT, AST and Alkaline Phosphatase
Description: Alanine aminotransferase [ALT], aspartate aminotransferase [AST], and alkaline phosphatase in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of Units per Liter (U/L)
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- SOV2012-F1-treated, Observed; SOV2012-F1-treated, Change From Baseline: Patients treated with SOV2012-F1, starting daily dose in MRS-TU-2019EXT is 400 mg - (200 mg with morning meal and 200 mg with evening meal). Dosing is titrated up to a maximum of 800 mg SOV2012-F1 per day (400 mg in the morning with morning meal and 400 mg in the evening with evening meal) or down to a minimum of 100 mg SOV2012-F1 per day (100 mg with morning meal) based on plasma T after 14 and 42 days of treatment. Patients could be titrated to final daily dose levels of 100 mg, 200 mg (100 mg twice daily), 400 mg (200 mg twice daily), 600 mg (300 mg twice daily) or 800 mg (400 mg twice daily). All doses taken with meals.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU) in 100 mg, 150 mg and 200 mg strengths.
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
U/L
  Alkaline Phosphatase, Baseline | 72.5 (22.90) | 0 (0)
  Alkaline Phosphatase, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Alkaline Phosphatase, Visit 12E - Day 90E | 70.4 (50.29) | -2.2 (33.68)
  Alkaline Phosphatase, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Alkaline Phosphatase, Visit 16E - EOT Day 180E | 65.0 (18.43) | -5.7 (10.60)
  Alanine Aminotransferase (ALT), Baseline | 32.0 (15.15) | 0 (0)
  Alanine Aminotransferase (ALT), Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Alanine Aminotransferase (ALT), Visit 12E - Day 90E | 26.5 (12.10) | -5.1 (13.37)
  Alanine Aminotransferase (ALT), Visit 16E - Day 180E: number analyzed (Participants) | 134 | 134
  Alanine Aminotransferase (ALT), Visit 16E - Day 180E | 26.9 (14.18) | -4.2 (14.46)
  Aspartate Aminotransferase (AST), Baseline | 24.1 (13.48) | 0 (0)
  Aspartate Aminotransferase (AST), Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Aspartate Aminotransferase (AST), Visit 12E - Day 90E | 22.5 (9.36) | -1.4 (14.26)
  Aspartate Aminotransferase (AST), Visit 16E - Day 180E: number analyzed (Participants) | 134 | 134
  Aspartate Aminotransferase (AST), Visit 16E - Day 180E | 21.6 (8.73) | -1.9 (13.28)

15. Other Pre Specified Outcome: Observed and Change From Baseline in Hematology Parameters in Liver Function Tests
Description: Total bilirubin in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of mg/dL
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
mg/dL
  Bilirubin, Baseline | 0.441 (0.2053) | 0 (0)
  Bilirubin, Visit 12E - Day 90: number analyzed (Participants) | 143 | 143
  Bilirubin, Visit 12E - Day 90 | 0.361 (0.1976) | -0.077 (0.1629)
  Bilirubin, Visit 16E - EOYDay 180: number analyzed (Participants) | 134 | 134
  Bilirubin, Visit 16E - EOYDay 180 | 0.431 (0.2383) | -0.004 (0.1863)

16. Other Pre Specified Outcome: Observed and Change From Baseline in Hematology Parameters (Hemoglobin) in SOV2012-F1 Treated Subjects During the Treatment Period.
Description: Hemoglobin in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of g/dL.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
g/dL
  Hemoglobin, Baseline: number analyzed (Participants) | 154 | 154
  Hemoglobin, Baseline | 14.72 (1.094) | 0 (0)
  Hemoglobin, Visit 12E - Day 90E: number analyzed (Participants) | 144 | 144
  Hemoglobin, Visit 12E - Day 90E | 15.13 (1.488) | 0.41 (1.082)
  Hemoglobin, Visit 16E - EOT Day 180E: number analyzed (Participants) | 134 | 134
  Hemoglobin, Visit 16E - EOT Day 180E | 15.19 (1.490) | 0.48 (1.068)

17. Other Pre Specified Outcome: Observed and Change From Baseline in Hormone Levels.
Description: Luteinizing hormone [LH] and follicle-stimulating hormone [FSH] in SOV2012-F1 treated subjects during the treatment period, measurement units of mIU/mL.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
mIU/mL
  Luteinizing Hormone, Baseline | 5.91 (4.119) | 0 (0)
  Luteinizing Hormone, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Luteinizing Hormone, Visit 12E - Day 90E | 2.13 (2.534) | -3.71 (4.410)
  Luteinizing Hormone, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Luteinizing Hormone, Visit 16E - EOT Day 180E | 2.39 (2.821) | -3.37 (4.342)
  Follicle Stimulating Hormone, Baseline | 5.83 (4.890) | 0 (0)
  Follicle Stimulating Hormone, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Follicle Stimulating Hormone, Visit 12E - Day 90E | 2.47 (3.037) | -3.28 (4.506)
  Follicle Stimulating Hormone, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Follicle Stimulating Hormone, Visit 16E - EOT Day 180E | 2.52 (3.073) | -3.19 (4.457)

18. Other Pre Specified Outcome: Observed and Change From Baseline in Hormone Levels for SHBG.
Description: Sex hormone-binding globulin [SHBG] in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of nmol/L.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
nmol/L
  Sex Hormone Binding Globulin, Baseline | 28.81 (14.193) | 0 (0)
  Sex Hormone Binding Globulin, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Sex Hormone Binding Globulin, Visit 12E - Day 90E | 20.30 (12.254) | -8.53 (7.901)
  Sex Hormone Binding Globulin, Visit 16E - EOT Day 180E: number analyzed (Participants) | 134 | 134
  Sex Hormone Binding Globulin, Visit 16E - EOT Day 180E | 18.97 (11.385) | -10.45 (8.630)

19. Other Pre Specified Outcome: Observed and Change From Baseline in Thyrotropin
Description: Thyroid stimulating hormone [TSH] in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of mU/L.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
mU/L
  Thyrotropin, Baseline | 3.014 (6.8492) | 0 (0)
  Thyrotropin, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Thyrotropin, Visit 12E - Day 90E | 2.985 (3.9809) | -0.101 (5.9459)
  Thyrotropin, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Thyrotropin, Visit 16E - EOT Day 180E | 2.263 (1.2560) | 0.003 (1.0863)

20. Other Pre Specified Outcome: Observed and Change From Baseline in Lipid Profiles in SOV2012-F1 Treated Subjects During the Treatment Period.
Description: Lipid profiles (high and low-density lipoproteins, total cholesterol, triglycerides) in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of mg/dL.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
mg/dL
  Cholesterol, Baseline | 186.4 (38.38) | 0 (0)
  Cholesterol, Visit 12E - Day 90E: number analyzed (Participants) | 144 | 144
  Cholesterol, Visit 12E - Day 90E | 171.7 (40.52) | -14.5 (31.69)
  Cholesterol, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Cholesterol, Visit 16E - EOT Day 180E | 176.2 (41.62) | -11.1 (30.50)
  HDL Cholesterol, Baseline | 45.3 (11.94) | 0 (0)
  HDL Cholesterol, Visit 12E - Day 90E: number analyzed (Participants) | 144 | 144
  HDL Cholesterol, Visit 12E - Day 90E | 37.2 (9.74) | -7.8 (7.75)
  HDL Cholesterol, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  HDL Cholesterol, Visit 16E - EOT Day 180E | 38.2 (10.37) | -6.9 (8.70)
  LDL Cholesterol, Baseline | 120.8 (35.85) | 0 (0)
  LDL Cholesterol, Visit 12E - Day 90E: number analyzed (Participants) | 144 | 144
  LDL Cholesterol, Visit 12E - Day 90E | 113.4 (37.52) | -7.8 (27.57)
  LDL Cholesterol, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  LDL Cholesterol, Visit 16E - EOT Day 180E | 117.7 (38.20) | -4.0 (29.14)
  Triglycerides, Baseline | 179.3 (123.60) | 0 (0)
  Triglycerides, Visit 12E - Day 90E: number analyzed (Participants) | 144 | 144
  Triglycerides, Visit 12E - Day 90E | 158.9 (83.79) | -16.7 (101.61)
  Triglycerides, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Triglycerides, Visit 16E - EOT Day 180E | 160.1 (102.90) | -18.6 (106.48)

21. Other Pre Specified Outcome: Observed and Change From Baseline in Serum Prostate-specific Antigen (PSA) in SOV2012-F1 Treated Subjects During the Treatment Period.
Description: Serum prostate-specific antigen (PSA) in SOV2012-F1 treated subjects were assessed during the treatment period, measurement units of ng/mL.
Time Frame: 90 and 180 days
Population: Extension Treated Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOV2012-F1-treated, Observed | SOV2012-F1-treated, Change From Baseline
Number analyzed (Participants) | 155 | 155
ng/mL
  Prostate Specific Antigen, Baseline | 0.98 (0.651) | 0 (0)
  Prostate Specific Antigen, Visit 12E - Day 90E: number analyzed (Participants) | 143 | 143
  Prostate Specific Antigen, Visit 12E - Day 90E | 1.10 (0.719) | 0.15 (0.309)
  Prostate Specific Antigen, Visit 16E - EOT Day 180E: number analyzed (Participants) | 135 | 135
  Prostate Specific Antigen, Visit 16E - EOT Day 180E | 1.09 (0.743) | 0.15 (0.443)

ADVERSE EVENTS:
Time Frame: 180 days
Description: All-Cause Mortality includes all causes; Serious Adverse events includes all causes; Other Adverse Events category includes only AE's judged by clinical investigators to have been treatment-related.
Arm/Group | SOV2012-F1-treated
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 2/155
Other Adverse Events (participants affected / at risk) | 30/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOV2012-F1-treated (N=155)
Atrial fibrillation (Cardiac disorders) | 1 (1) — Event judged not treatment related by investigator.
Diverticular perforation (Gastrointestinal disorders) | 1 (1) — Event judged not treatment related by investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOV2012-F1-treated (N=155)
Hypertension (Vascular disorders) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 8 (8)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5)
Influenza (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3)
Hemoglobin increased (Investigations) | 3 (3) — Event judged as treatment related by investigator.
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04467697/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04467697/SAP_001.pdf